CLINICAL TRIAL: NCT06380894
Title: Virtual Reality Cognitive Training for Mild Cognitive Impairment - A Pilot Feasibility Study
Brief Title: Virtual Reality Cognitive Training for Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2020/2239
Record Dates: First submitted 2024-04-10; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Cognitive Training (Experimental): The program consisted of two components: (1) psychoeducation on cognitive functioning and ways to maintain cognitive health, (2) VR multi-domain cognitive training tasks that target cognitive domains of attention, memory, and executive functioning.
  Interventions: Device: Virtual Reality Cognitive Training
- Active Control Group (Active Comparator): Participants who were assigned to the active control group were provided treatment-as-usual, which included: (1) psychoeducation on MCI, cognitive functioning, and compensatory strategies, and (2) brain training cognitive stimulation booklet which consisted of weekly homework activities focusing on attention, memory, and executive functioning. Control participants were reviewed for 3 sessions monthly to follow up on their progress on the cognitive stimulation activity booklet.
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Device: Virtual Reality Cognitive Training — Participants who were assigned to the VRCT intervention group underwent 60 minutes of weekly VRCT sessions over a 10-week intervention period. The program consisted of two components: (1) psychoeducation on cognitive functioning and ways to maintain cognitive health, (2) VR multi-domain cognitive training tasks that target cognitive domains of attention, memory, and executive functioning.
  The VR experiences were administered through a head-mounted Oculus Go Screen V7. The VR system runs on a software developed by Dancing Mind Pte Ltd. The software specifications and service provided by Dancing Mind Pte Ltd include: MindGym System Functions: System Setup (Processor Setup, Password Changing etc) and Data Centre (Memory Care Therapy Data Analytics Report Querying and Printing Functions). The MindGym cognitive training content was developed based on the Singaporean culture, with visual stimuli reflecting familiar local environments.
  Arms: Virtual Reality Cognitive Training
Behavioral: Active Control — Participants who were assigned to the active control group were provided treatment-as-usual, which included: (1) psychoeducation on MCI, cognitive functioning, and compensatory strategies, and (2) brain training cognitive stimulation booklet which consisted of weekly homework activities focusing on attention, memory, and executive functioning. Control participants were reviewed for 3 sessions monthly to follow up on their progress on the cognitive stimulation activity booklet.
  Arms: Active Control Group

SUMMARY:
This study aims to assess the feasibility and efficacy of a 10-weekly multi-domain VRCT program on the cognitive function (i.e. attention, memory, and executive functioning) of older adults with MCI.

DETAILED DESCRIPTION:
This study employed a pilot feasibility parallel design approach. Participants were randomly assigned to either the VRCT intervention group or the active control group. The outcome assessor was blinded. Participants were recruited from outpatient clinics in Changi General Hospital, Singapore. They were referred by treating geriatricians and psycho-geriatricians.

ELIGIBILITY:
Inclusion Criteria:

* aged 65-85
* diagnosis of MCI by a clinician in accordance to Petersen's criteria
* MMSE ≥ 23
* ability to see and hear
* ability to read and write in either English or Mandarin

Exclusion Criteria:

* diagnosed with a primary other neurocognitive disorder
* diagnosed with major psychiatric illness such as major depressive disorder or anxiety disorder, severe visual or auditory impairment
* diagnosed with serious medical illnesses including acute or severe asthma, severe or unstable cardiovascular disease, active gastric ulcer, severe liver disease or severe renal disease.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Memory Performance on the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) subtests at Week 11 | Baseline and Week 11
  The RBANS is a comprehensive neuropsychological battery that has been validated with local norms in Singapore. Its subtests of List Learning, List Recall and List Recognition measures verbal memory while Picture Copy and Picture Recall measures visual memory. It is administered by trained clinical research coordinators and scored by neuropsychologists. Raw scores of each subtests are compared.
Change from Baseline in Attention Performance on the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) subtest at Week 11 | Baseline and Week 11
  The RBANS is a comprehensive neuropsychological battery that has been validated with local norms in Singapore. Its subtest of Digit Span measures attention. It is administered by trained clinical research coordinators and scored by neuropsychologists. Raw scores of the Digit Span subtest is compared.
Change from Baseline in Attention Performance on the Colour Trails Test 1 at Week 11 | Baseline and Week 11
  The Colour Trails Test 1 requires the respondent to connect circles in an ascending numbered sequence. Time taken to complete each part of the CTT is recorded in seconds.
Change from Baseline in Executive Function Performance on the Frontal Assessment Battery (FAB) at Week 11 | Baseline and Week 11
  The FAB is a short screening tests used to evaluate executive function. Its components consist of S-word generation, similarities, Luria's test, grasp reflex, and the Go-No-Go test. The sum of the sub-scores from each of the six components are added up to generate total score out of 18.
Change from Baseline in Executive Function Performance on the Colour Trails Test 2 at Week 11 | Baseline and Week 11
  The FAB is a short screening tests used to evaluate executive function. Its components consist of S-word generation, similarities, Luria's test, grasp reflex, and the Go-No-Go test. The sum of the sub-scores from each of the six components are added up to generate total score out of 18.

CONTACTS AND LOCATIONS:
Overall Officials: Zhong Jie Zaylea Kua, MPsychClin, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-27): https://cdn.clinicaltrials.gov/large-docs/94/NCT06380894/Prot_SAP_000.pdf